CLINICAL TRIAL: NCT06467656
Title: The UBC Long-distance Triathlon Adaptation Study
Acronym: ULTRA
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of British Columbia (Other)
Responsible Party: Principal Investigator, Robert Shave, Professor, University of British Columbia
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: H24-00882
Record Dates: First submitted 2024-05-22; First posted 2024-06-21 (Actual); Last update posted 2025-04-04 (Actual); Status verified 2025-04

CONDITIONS: Healthy Participants
Keywords: Exercise; Endurance training; Cardiorespiratory fitness; Cardiovascular; Respiratory; Vascular; Immune; Microbiome; Psychology; Performance; Biological Sex Differences
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: This will be a parallel group, non-randomized study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exercise Intervention (Experimental): Participants will engage in 12 months of individualized endurance-training (swimming, cycling and running) and 9 months of supplemental strengthening exercises. Exercise prescriptions will be provided to participants weekly via an app (TrainingPeaks). Sessions will vary in length from 30 min to 8 hours throughout the program.
  Interventions: Other: Individualized, periodized endurance training for ultra-endurance triathlon.
- Time-Aligned Control (Active Comparator): Participants in the control arm will continue to live their lives exactly as they would if they were not enrolled in a study to allow evaluation of natural biological changes that occur across 12-months of free-living.
  Interventions: Other: Time-Aligned Control

INTERVENTIONS:
Other: Individualized, periodized endurance training for ultra-endurance triathlon. — Endurance exercise consisting of swimming, cycling and running training for a minimum of 3 hours /week up to a maximum of 20 hours/week with regular rest days and intensities being fluctuated throughout the program to optimize training stimulus and adaptation. Strengthening exercises to complement the aerobic training, enhance conditioning and prevent injury will also be performed 1-2 hours/week for the first 9-months of the program.
  Arms: Exercise Intervention
Other: Time-Aligned Control — Participants will receive no specific intervention and will continue to live their lives as if they were not in a study.
  Arms: Time-Aligned Control

SUMMARY:
The purpose of this study is to investigate the effect of 12-months of individualized endurance-training (swimming, cycling and running) on physiological and psychological adaptations in exercise naïve individuals. Due to the potential seasonal changes that naturally occur in individuals across a year (even without training) the investigators will also compare the exercise-trained group to a time-aligned control group.

DETAILED DESCRIPTION:
Endurance training is well-accepted to lead to numerous positive physiological and psychological adaptations. However, many of the previous studies examining the benefits of endurance exercise on the human body have: 1) compared athletes with non-athletes using a cross-sectional design, 2) have employed training studies that are relatively short (e.g. weeks to months) in duration, 3) have primarily focused on male participants and not examined potential sex-differences, and 4) have not specifically recruited exercise naïve participants, as often participants are already engaged in ongoing recreational or competitive activities at the time of recruitment. As such, we have a limited understanding of the true time-course of adaptations that occur in exercise naïve individuals in response to training, or how physiological and psychological adaptations change beyond 4-6 months, and whether there are sex-specific differences in these adaptations.

This study is primarily designed to determine the time-course of adaptation and remodeling in females and males across multiple different physiological systems (i.e. cardiac, vascular, metabolic, respiratory, immune, and microbiome) and psychological measures at rest and in response to a range of provocations.

Forty healthy exercise-training naïve individuals (20 females: 20 males) will perform 12-months of individually prescribed, endurance training (including supplementary strengthening exercise for conditioning and injury prevention) designed to prepare participants for an ultra-endurance triathlon. A time-aligned control group of 20 healthy exercise-training naïve individuals (10 females: 10 males) will also be recruited to determine the natural change that occurs in each system across a year. Outcomes will be assessed at baseline, 3 months, 6 months and 12 months. Additionally, cardiovascular outcomes will also be assessed at 1 month and immune outcomes will be repeated at 3 months post intervention (15 months).

ELIGIBILITY:
Inclusion Criteria: Exercise Intervention Group

* Aged 19-39 years
* Non-smoker (quit >6 months)
* Able to swim >100 meters without stopping
* Have access to, or willingness, to obtain a road bicycle
* Are willing to commit to the research assessments and prescribed training program
* Currently performing <120 minutes of structured endurance training per week
* Premenopausal

Inclusion Criteria: Control Group

* Aged 19-39 years
* Non-smoker (quit >6 months)
* Are willing to commit to the research assessments
* Currently performing <120 minutes of structured endurance training per week
* Premenopausal

Exclusion Criteria: Exercise Intervention Group and Control Group:

* History of heart disease
* History of lung disease (not including controlled asthma)
* History of metabolic disease
* History of cancer
* Chronic inflammatory conditions
* Blood pressure > 140/90 mmHg
* Chronic antibiotic, antiviral, antimicrobial, non-steroidal anti-inflammatory drugs (NSAIDs) and antihistamine use
* Are a regular (more than 1/week) cannabis user
* Consume alcohol regularly: more than 6 standard drinks per week (e.g.14-20 ounces of beer and 5-8 ounces of wine)
* Have previously completed structured endurance exercise training for an extended period of time (such as training for a triathlon or running race)
* Have previously participated in competitive team sports with an aerobic component (e.g. soccer, basketball, rugby, field hockey) and sport-specific training (e.g. hockey, football) >3 times per week within the previous 5 years
* Have prior experience of heavy structured resistance training >3x/week within the last 2 years
* BMI>32 kg/m2 or <20 kg/m2
* Pregnancy within 12 months, or planning to become pregnant within the next 12 months
* Currently breast feeding (or having stopped within 6 months)
* Planning to be away from the Okanagan area for an extended period over the duration of the study

Ages: 19 Years to 39 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-06-20 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen consumption (VO2max). | 12 Months
  The change in VO2max from baseline to 12 months of exercise training.

SECONDARY OUTCOMES:
Time-course of change in VO2max. | 3, 6, and 12 months
  The time-course of change in VO2max from baseline to 3, 6, and 12 months of exercise training.
Time-course of change in resting left ventricular structure. | 1, 3, 6, and 12 months
  The time-course of change in left ventricular end-diastolic volume (via transthoracic echocardiography) at rest from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in left ventricular structure during exercise. | 1, 3, 6, and 12 months
  The time-course of change in left ventricular end-diastolic volume (via transthoracic echocardiography) during acute exercise from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in left ventricular structure with volume loading. | 1, 3, 6, and 12 months
  The time-course of change in left ventricular end-diastolic volume (via transthoracic echocardiography) in response to head down tilt from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in ventricular diameter to wall thickness | 1, 3, 6, and 12 months
  The time-course of change in the ratio of ventricular diameter to ventricular wall thickness (via transthoracic echocardiography) at rest from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in left ventricular mass | 1, 3, 6, and 12 months
  The time-course of change in left ventricular mass (via transthoracic echocardiography) at rest from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in resting right ventricular structure. | 1, 3, 6, and 12 months
  The time-course of change in right ventricular area (via transthoracic echocardiography) at rest, from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in right ventricular structure during exercise. | 1, 3, 6, and 12 months
  The time-course of change in right ventricular area (via transthoracic echocardiography) in response to exercise from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in right ventricular structure with volume loading. | 1, 3, 6, and 12 months
  The time-course of change in right ventricular area (via transthoracic echocardiography) in response to head-down tilt from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in resting left atrial structure. | 1, 3, 6, and 12 months
  The time-course of change in resting left atrial phasic volumes (via transthoracic echocardiography) at rest from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in left atrial structure during exercise. | 1, 3, 6, and 12 months
  The time-course of change in left atrial phasic volumes (via transthoracic echocardiography) in response to exercise from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in left atrial structure with volume loading. | 1, 3, 6, and 12 months
  The time-course of change in left atrial phasic volumes (via transthoracic echocardiography) in response to head-down tilt from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in resting left ventricular function. | 1, 3, 6, and 12 months
  The time-course of change in left ventricular stroke volume (via transthoracic echocardiography) at rest from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in left ventricular function during exercise. | 1, 3, 6, and 12 months
  The time-course of change in left ventricular stroke volume (via transthoracic echocardiography) in response to acute exercise from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in left ventricular function with volume loading. | 1, 3, 6, and 12 months
  The time-course of change in left ventricular stroke volume (via transthoracic echocardiography) in response to head-down tilt from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in resting left ventricular diastolic function. | 1, 3, 6, and 12 months
  The time-course of change in the ratio of early to late left ventricular filling velocities (via transthoracic echocardiography) at rest from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in resting right ventricular function. | 1, 3, 6, and 12 months
  The time-course of change in right ventricular fractional area change (via transthoracic echocardiography) at rest, from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in right ventricular function during exercise. | 1, 3, 6, and 12 months
  The time-course of change in right ventricular fractional area change (via transthoracic echocardiography) in response to acute exercise, from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in right ventricular function with volume loading. | 1, 3, 6, and 12 months
  The time-course of change in right ventricular fractional area change (via transthoracic echocardiography) in response to head down tilt, from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in resting right ventricular strain. | 1, 3, 6, and 12 months
  The time-course of change in right ventricular longitudinal strain (via transthoracic echocardiography) at rest, from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in right ventricular strain during exercise. | 1, 3, 6, and 12 months
  The time-course of change in right ventricular longitudinal strain (via transthoracic echocardiography) in response to acute exercise, from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in right ventricular strain with volume loading. | 1, 3, 6, and 12 months
  The time-course of change in right ventricular longitudinal strain (via transthoracic echocardiography) in response to head down tilt, from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in resting left-atrial strain | 1, 3, 6, and 12 months
  The time-course of change in left atrial phasic strain (via transthoracic echocardiography) at rest from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in left-atrial strain during exercise. | 1, 3, 6, and 12 months
  The time-course of change in left atrial phasic strain (via transthoracic echocardiography) in response to acute exercise, from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in in left-atrial strain with volume loading. | 1, 3, 6, and 12 months
  The time-course of change in left atrial phasic strain (via transthoracic echocardiography) in response to head down tilt, from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in p-wave duration. | 1, 3, 6, and 12 months
  The time-course of change in p wave duration (by 12-lead electrocardiography and signal-averaged electrocardiography) at rest from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in p-wave amplitude | 1, 3, 6, and 12 months
  The time-course of change in p wave amplitude (by 12-lead electrocardiography and signal-averaged electrocardiography) at rest from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Time-course of change in p wave root mean square average | 1, 3, 6, and 12 months
  The time-course of change in p wave root mean square voltage (by signal-averaged electrocardiography) at rest from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Relationships between changes in cardiac electrical activity and left atrial volume. | 1, 3, 6, and 12 months
  The relationship between p wave duration (by 12-lead electrocardiography and signal-averaged electrocardiography), amplitude (by 12-lead electrocardiography and signal-averaged electrocardiography) and root mean square voltage (by signalaveraged electrocardiography) with left atrial volume (via transthoracic echocardiography) from baseline to 3, 6 and 12 months of exercise training.
Time-course of change in blood volume. | 1, 3, 6, and 12 months
  The time-course of change in blood volume (using the carbon monoxide re-breathe technique) from baseline to 1, 3, 6 and 12 months of exercise-training and compared to the change in the time-aligned control group.
Relationship between changes in blood volume and cardiac structure | 1, 3, 6, and 12 months
  The relationship between changes in blood volume and changes in cardiac structure (left ventricular end diastolic volume, ratio of ventricular diameter to ventricular wall thickness, ventricular mass, right ventricular area, left atrial volume; via transthoracic echocardiography) and function (stroke volume, right ventricular fractional area change, ratio of early to late left ventricular filling velocities, left ventricular longitudinal strain and left atrial strain; via transthoracic echocardiography) from baseline to 1, 3, 6 and 12 months of exercise training.
Time-course of change in resting upper body vascular structure. | 1, 3, 6, and 12 months
  The time-course of change in upper body macrovascular structure by resting brachial artery diameter.
Time-course of change in upper body vascular structure. | 1, 3, 6, and 12 months
  The time-course of change in upper body macrovascular structure by maximal brachial artery diameter following ischemic hand-grip from baseline to 1,3, 6 and 12 months of exercise training.
Time-course of change in resting lower body vascular structure. | 1, 3, 6, and 12 months
  The time-course of change in lower body macrovascular structure by resting superficial femoral artery diameter.
Time-course of change in upper body microvascular structure. | 1, 3, 6, and 12 months
  The time-course of change in upper body microvascular structure from the maximal hyperemic response to hand-grip ischemic exercise from baseline to 1,3, 6 and 12 months of exercise training.
Time-course of change in upper body vascular function. | 1, 3, 6, and 12 months
  The time-course of change in upper body macrovascular function by brachial artery flow mediated dilation from baseline to 1,3,6 and 12 months of exercise training.
Time-course of change in lower body vascular function. | 1, 3, 6, and 12 months
  The time-course of change in lower body macrovascular function by superficial femoral artery flow mediated dilation from baseline to 1,3,6 and 12 months of exercise training.
Time-course of change in upper body microvascular function | 1, 3, 6, and 12 months
  The time-course of change in upper body microvascular function by the brachial artery reactive hyperemia response from baseline to 1,3,6 and 12 months of exercise training.
Time-course of change in lower body microvascular function. | 1, 3, 6, and 12 months
  The time-course of change in lower body microvascular function by the superficial femoral artery reactive hyperemia response from baseline to 1,3,6 and 12 months of exercise training.
Time-course of change in arterial stiffness. | 1, 3, 6, and 12 months
  Central arterial stiffness (carotid-femoral pulse wave velocity) from baseline to 1,3,6 and 12 months of exercise training.
Change in exercising ventilatory reserve | 12 months
  Change in ventilatory reserve (maximum ventilation / ventilatory capacity) from baseline to 12 months of exercise training.
Change in expiratory flow limitation. | 12 months
  Change in expiratory flow limitations (% overlap of the exercise flow-volume loop at max exercise with the maximum flow-volume envelope) from baseline to 12 months of exercise training.
Change in work of breathing. | 12 months
  Change in total work of breathing (measured as the combination of inspiratory resistive, inspiratory elastic, and expiratory resistive work of breathing assessed by modified Campbell diagram) at intensity-matched exercise from baseline to 12 months of exercise training.
Change in ventilatory efficiency. | 12 months
  Change in ventilatory efficiency (assessed by VE-VCO2 slope during graded exercise) from baseline to 12 months of exercise training.
Change in lung volume. | 12 months
  Change in operational lung volumes (assessed via IC maneuvers) during intensity-matched exercise from baseline to 12 months of exercise training.
Change in dyspnea. | 12 months
  Change in dyspnea (assessed via modified Borg scale) during intensity-matched exercise from baseline to 12 months of exercise training.
Time course of change in exercising ventilatory reserve | 3, 6, and 12 months
  Time course of change in ventilatory reserve (maximum ventilation / ventilatory capacity) from baseline to 3, 6, and 12 months of exercise training.
Time course of change in expiratory flow limitation. | 3, 6, and 12 months
  Time course of change in the expiratory flow limitation (% overlap of the exercise flow-volume loop at max exercise with the maximum flow-volume envelope) from baseline to 3, 6, and 12 months of exercise training.
Time course of change in work of breathing. | 3, 6, and 12 months
  Time course of change in total work of breathing (measured as the combination of inspiratory resistive, inspiratory elastic, and expiratory resistive work of breathing assessed by modified Campbell diagram) at intensity-matched exercise from baseline to 12 months of exercise training.
Time course of change in ventilatory efficiency. | 3, 6, and 12 months
  Time course of change in ventilatory efficiency (assessed by VE-VCO2 slope during graded exercise) from baseline to 12 months of exercise training.
Time course of change in lung volume. | 3, 6, and 12 months
  Time course of change in operational lung volumes (assessed via IC maneuvers) during intensity-matched exercise from baseline to 12 months of exercise training.
Time course of change in dyspnea. | 3, 6, and 12 months
  Time course of change in dyspnea (assessed via modified Borg scale) during intensity-matched exercise from baseline to 12 months of exercise training.
Time course of change in chemoreflex sensitivity. | 3, 6, and 12 months
  Time course of change in chemoreflex sensitivity (ventilatory response to changes in inspired CO2 and O2) from baseline to 3, 6, and 12 months of exercise training.
Gut microbiome composition and diversity. | 1,3, 6, and 12 months
  The time course of change in gut microbiome composition and diversity (microbial alpha and beta diversity by 16S rRNA gene sequencing or shotgun metagenomic sequencing), circulating metabolites [plasma short-chain fatty acids (SCFA) and trimethylamine N-oxide (TMAO) levels], and markers of inflammation (fecal calprotectin and plasma cytokines via ELISA) and gut permeability [plasma lipopolysaccharide (LPS) via ELISA] from baseline to 1, 3, 6 and 12 months of exercise training.
Relationships between gut microbiome and exercise performance | 1,3, 6, and 12 months
  The relationship (as assessed through regression analyses) between changes in the gut microbiome with improvements in exercise performance from baseline to 1, 3, 6 and 12 months of exercise training.
Relationships between gut microbiome and cardio metabolic health | 1,3, 6, and 12 months
  The relationship (as assessed through regression analyses) between changes in the gut microbiome, microbiome-driven metabolites (SCFA and TMAO), markers of inflammation (fecal calprotectin and plasma cytokines), and indices of gut permeability (plasma LPS) relevant to cardiometabolic health from baseline to 1,3, 6 and 12 months of exercise training.
Innate immune reprogramming. | 12 months
  The change in epigenomic landscape and cell function (e.g., cytokine production, phagocytosis) of circulating monocytes from baseline to 12 months of exercise training and compared to the change in the time-aligned control group.
Innate immune memory. | 15 months
  The change in epigenomic landscape and cell function (e.g., cytokine production, phagocytosis) of circulating monocytes from 12-month exercise training to 3 months post exercise cessation.
Affective response. | 12 months
  The time course of changes in affective responses specifically exercise valence and arousal that people experience while exercising using a 1-item affect grid from baseline to 12 months and compared to the change in the time-aligned control group.
Affective processing. | 12 months
  The time course of changes in affective processing (i.e pleasure-displeasure, energy-tired, calmness-tension, attraction-antipathy, pride/honour-guilt/shame, empowerment-damage) that people experience from baseline to 12 months and compared to the change in the time-aligned control group.
Relationships between affective responses, affective processing and other exercise and psychological variables. | 12 months
  The relationships (as assessed through regression analyses) between affective responses, affective processing, incidental affect, exercise identity, competence, and adherence behaviours as well as cardiopulmonary fitness.
Time course of change in blood lactate. | 3, 6, and 12 months
  Change in blood lactate (fingertip lactate) during sustained moderate-high intensity exercise from baseline to 3, 6, and 12 months of exercise training.
Time course of change in heart rate. | 3, 6, and 12 months
  Change in heart rate (telemetry) during sustained moderate-high intensity exercise from baseline to 3, 6, and 12 months of exercise training.
Time course of change in perceived exertion. | 3, 6, and 12 months
  Change in rating of perceived exertion (modified Borg scale) during sustained moderate-high intensity exercise from baseline to 3, 6, and 12 months of exercise
Sex-difference in physiological adaptation. | 1,3, 6, 12 and 15 months where applicable
  Sex-differences in the time course of change in physiological parameters associated with the primary and secondary outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Shave, PhD, Principal Investigator — University of British Columbia
Locations (1):
- University of British Columbia, Kelowna, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: Yes
Requests for deidentified individual participant data can be made 6 months following publication. Deidentified individual participant data reported in manuscripts will be shared but may need a data sharing agreement in place between UBC and the institution of the requester.
Time Frame: Ongoing from 6 months after publication